CLINICAL TRIAL: NCT03333044
Title: Diabetes Management Intervention For South Asians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-01479; U54MD000538-15 (NIH)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: HbA1c; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW-Led Health Coaching (Experimental): Participants in the treatment group will be randomized to receive the CHW group education session intervention in either the first or second round.
  Interventions: Behavioral: Community Health Worker (CHW)-Led Health Coaching; Other: EHR-Embedded Alerts
- Wait-List Control (No Intervention): Participants in the wait-list control group will be receive care as usual during the first round for data abstraction and offered CHW group education sessions during the second round as a point of service (i.e., not for research purposes).

INTERVENTIONS:
Behavioral: Community Health Worker (CHW)-Led Health Coaching — CHW intervention includes a protocol that consists of 5 monthly 90-minute group health education sessions, providing the tools and strategies to manage diabetes.
  Arms: CHW-Led Health Coaching
Other: EHR-Embedded Alerts — An electronic health record (EHR) intervention for primary care providers (PCPs) utilizing embedded alerts to identify South Asian patients with uncontrolled diabetes.
  Arms: CHW-Led Health Coaching

SUMMARY:
The goal of this study is to evaluate the effectiveness and implementation process of a multi-level, integrated intervention to decrease HbA1c among South Asians with uncontrolled diabetes, including four components: 1) an EHR-based registry function to increase identification of South Asian patients with uncontrolled diabetes; 2) CHW-led health coaching of registered patients to promote health behavior change; 3) HIT-enabled and CHW-facilitated identification and referral to culturally relevant community resources for patients; and 4) HIT-enabled care coordination between the CHW and other members of the healthcare team.

ELIGIBILITY:
Inclusion Criteria:

* South Asian ethnicity (identified through a race and language code available in the EHR);
* an appointment with a physician for routine non-emergent primary care in the last 12 months
* diagnosis of diabetes
* an HbA1c reading of >7 in the last 12 months

Exclusion Criteria:

* Pregnant women and visits to obstetrician/gynecologist are excluded from the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- One Park Avenue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: AFTER FINAL DATA COLLECTION AND FOLLOWING PUBLICATION OF MAIN FINDINGS MANUSCRIPT
Access Criteria: Researchers who provide a methodologically sound proposal. Requests should be directed to Shinu.Mammen@nyulangone.org To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Mohsin F, Wyatt L, Belli H, Ali S, Onakomaiya D, Misra S, Yusuf Y, Mammen S, Zanowiak J, Hussain S, Zafar H, Lim S, Islam N, Ahmed N. Diabetes distress among immigrants of south Asian descent living in New York City: baseline results from the DREAM randomized control trial. BMC Public Health. 2025 Feb 2;25(1):422. doi: 10.1186/s12889-025-21535-8. PMID 39894868
- [Derived] Hu L, Wyatt LC, Mohsin F, Lim S, Zanowiak J, Mammen S, Hussain S, Ali SH, Onakomaiya D, Belli HM, Aifah A, Islam NS. Characterizing Technology Use and Preferences for Health Communication in South Asian Immigrants With Prediabetes or Diabetes: Cross-Sectional Descriptive Study. JMIR Form Res. 2024 Apr 26;8:e52687. doi: 10.2196/52687. PMID 38669062
- [Derived] Mohsin F, Wyatt L, Belli H, Ali S, Onakomaiya D, Misra S, Yusuf Y, Mammen S, Zanowiak J, Hussain S, Zafar H, Lim S, Islam N, Ahmed N. The Prevalence and Correlates of Diabetes Distress among South Asians Living in New York City (NYC): Baseline Results from a Randomized Trial. Res Sq [Preprint]. 2023 Jun 8:rs.3.rs-2806895. doi: 10.21203/rs.3.rs-2806895/v1. PMID 37333263
- [Derived] Lim S, Wyatt LC, Mammen S, Zanowiak JM, Mohaimin S, Troxel AB, Lindau ST, Gold HT, Shelley D, Trinh-Shevrin C, Islam NS. Implementation of a multi-level community-clinical linkage intervention to improve glycemic control among south Asian patients with uncontrolled diabetes: study protocol of the DREAM initiative. BMC Endocr Disord. 2021 Nov 23;21(1):233. doi: 10.1186/s12902-021-00885-5. PMID 34814899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Primary care providers (PCPs) were not considered enrolled in this study.
Units Other Than Participants: Clinics
Groups:
- Waive 1 (10/2018-12/2019) Round 1 Jan-Jun 2019, Round 2 July-Dec 2019: All participants waitlisted during the Waive 1- Round 1 were randomized to the Waive 1 Wait-List Control group.
  During the first round (Jan-Jun 2019), participants received standard of care. During the second round (July-Dec 2019), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 1 received the intervention from Jan-Jun 2019 for Round 1; Round 2 participants received the intervention from July-Dec 2019.
- Waive 2 (10/2019-12/2020) Round 1 Jan-Jun 2020, Round 2 July-Dec 2020: All participants waitlisted during the Waive 2 - Round 1 were randomized to the Waive 2 Wait-List Control group.
  During the first round (Jan-Jun 2020), participants received standard of care. During the second round (July-Dec 2020), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 2 received the intervention from Jan-Jun 2020 for Round 1; Round 2 participants received the intervention from July-Dec 2020.
- Waive 3 (10/2020-12/2021) Round 1 Jan-Jun 2021, Round 2 July-Dec 2021: All participants waitlisted during the Waive 3 - Round 1 were randomized to the Waive 3 Wait-List Control group.
  During the first round (Jan-Jun 2021), participants received standard of care. During the second round (July-Dec 2021), all control participants were offered the full CHW group education sessions, though not for research purposes.
  Participants randomized to receive the intervention in Waive 3 received the intervention from Jan-Jun 2021 for Round 1; Round 2 participants received the intervention from July-Dec 2021.
Period: Overall Study
Arm/Group | Waive 1 (10/2018-12/2019) Round 1 Jan-Jun 2019, Round 2 July-Dec 2019 | Waive 2 (10/2019-12/2020) Round 1 Jan-Jun 2020, Round 2 July-Dec 2020 | Waive 3 (10/2020-12/2021) Round 1 Jan-Jun 2021, Round 2 July-Dec 2021
Started | 293; 7 Clinics | 314; 7 Clinics | 252; 5 Clinics
Participants Started Wait-List Control Round 1, CHW Round 2 | 146; 7 Clinics | 150; 7 Clinics | 123; 5 Clinics
Participants Completed Wait-List Control Round 1, CHW Round 2 | 146; 7 Clinics | 150; 7 Clinics | 123; 5 Clinics
Participants Started CHW Round 1, CHW Round 2 | 147; 7 Clinics | 164; 7 Clinics | 129; 5 Clinics
Participants Completed CHW Round 1, CHW Round 2 | 146; 7 Clinics | 150; 7 Clinics | 123; 5 Clinics
Completed | 292; 7 Clinics | 300; 7 Clinics | 246; 5 Clinics
Not Completed | 1; 0 Clinics | 14; 0 Clinics | 6; 0 Clinics
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 14 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait-List Control | CHW-Led Health Coaching | Total
Number analyzed (Participants) | 419 | 419 | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (9.7) | 55.1 (9.7) | 55.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 223 | 445
  Male | 197 | 196 | 393
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 419 | 419 | 838
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 419 | 419 | 838
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 419 | 419 | 838

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had at Least a 0.5% Reduction in HbA1c From Baseline 6 Months
Description: Measured via complete lipoprotein panel.
Time Frame: Baseline, Month 6
Measure: Number; unit: Percentage of participants
Arm/Group | Wait-List Control | CHW-Led Health Coaching
Number analyzed (Participants) | 196 | 219
Percentage of participants | 32.1 | 35.2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Wait-List Control | CHW-Led Health Coaching
All-Cause Mortality (participants affected / at risk) | 0/419 | 0/440
Serious Adverse Events (participants affected / at risk) | 0/419 | 0/440
Other Adverse Events (participants affected / at risk) | 0/419 | 0/440

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/44/NCT03333044/Prot_SAP_000.pdf